CLINICAL TRIAL: NCT02885831
Title: Early Abduction Splintage on Stable Hips in Infants With Developmental Dysplasia of the Hip : Improvement or Overtreatment ?
Brief Title: Early Abduction Splintage on Stable Hips in Infants With Developmental Dysplasia of the Hip
Acronym: BBH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: BBH (RB 16-057)
Record Dates: First submitted 2016-08-11; First posted 2016-09-01 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Congenital Hip Dysplasia
Keywords: Abduction splint; Pubo-femoral distance
MeSH Terms: conditions — Hip Dislocation, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A - Abduction splintage: Treatment by abduction splintage. Sonographic, clinical and radiographic surveillance. 45 patients.
  Interventions: Device: Abduction splintage
- B - Surveillance: No treatment by abduction splintage. Sonographic, clinical and radiographic surveillance. 45 patients

INTERVENTIONS:
Device: Abduction splintage — Treatment by abduction splintage 24 hours a day and 7 days a week, for 2 months.
  Other Names: Neut Supple Hip Abduction Cushion Without Bone
  Groups: A - Abduction splintage

SUMMARY:
The aim of this study is to prove the improvement of pubo-femoral distance by early abduction splintage in one-month-old infants with developmental dysplasia of the hip (with a clinical stable hip but an abnormal hip ultrasonography).

ELIGIBILITY:
Inclusion Criteria:

* Term infants
* Infants between 1 and 2 months of age at inclusion
* Clinically stable hip
* Pathological ultrasonography : pubo-femoral distance >6mm and bony rim percentage <50%
* Non objection of the family

Exclusion Criteria:

* Clinically unstable hip
* Normal ultrasonography
* Neuro-orthopedic disease
* Postural deformity of the pelvis
* Participation refusal

Ages: 1 Month to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants who underwent ultrasonographic screening for developmental dysplasia of the hip and are adressed to a paediatric orthopaedic surgeon at Brest University Hospital.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2016-12-08 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Normal or abnormal hip ultrasound | 2 months
  A normal or abnormal hip ultrasound will be base on two outcomes :
  * Pubo-femoral distance (ultrasonographic measurement) : distance between the pubic bone and the cartilaginous femoral head, considered as normal if lower than 6mm.
  * Bony rim percentage (ultrasonographic measurement) : percentage of the cartilaginous femoral head covered by the acetabular roof, considered as normal if higher than 50% (or equal to 50%).
  * Data of pubo-femoral distance and bony rim percentage will be pooled to determine if the ultrasound is normal or not for each patient. If one out of two is abnormal, ultrasound is considered abnormal. Statistics will be based on this qualitative value : normal or abnormal ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias THEPAUT, PhD, Principal Investigator — University Hospital, Brest
Locations (1):
- CHRU de Brest, Brest, France

REFERENCES:
- [Derived] Dwan K, Kirkham J, Paton RW, Morley E, Newton AW, Perry DC. Splinting for the non-operative management of developmental dysplasia of the hip (DDH) in children under six months of age. Cochrane Database Syst Rev. 2022 Oct 10;10(10):CD012717. doi: 10.1002/14651858.CD012717.pub2. PMID 36214650